CLINICAL TRIAL: NCT00406367
Title: Prospective, Double-blind, Placebo-controlled, Randomized, Multi-center Trial With an Open-label Extension Period to Investigate the Efficacy and Safety of incobotulinumtoxinA (Xeomin) in the Treatment of Blepharospasm
Brief Title: IncobotulinumtoxinA (Xeomin) Versus Placebo in the Treatment of Blepharospasm
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRZ 60201-0433
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Results first posted 2010-11-16 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Blepharospasm
MeSH Terms: conditions — Blepharospasm | interventions — incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- incobotulinumtoxinA (Xeomin) (Experimental): incobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kiloDalton), free from complexing proteins") powder for solution for injection dose (Main Period only): one injection session of solution, prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl), up to 50 Units per eye; Open-Label Extension Period: up to 5 injections, up to 50 Units per eye per injection session; Mode of administration: intramuscular injection
  Interventions: Drug: incobotulinumtoxinA (Xeomin)
- Placebo (Placebo Comparator): Placebo to incobotulinumtoxinA (Xeomin) powder for solution for injection dose (Main Period only): one injection session of solution, prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl), placebo volume corresponding to up to 50 Units per eye; Mode of administration: intramuscular injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: incobotulinumtoxinA (Xeomin) — incobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kiloDalton), free from complexing proteins") (active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection, up to 50 Units per eye; Mode of administration: intramuscular injection
  Arms: incobotulinumtoxinA (Xeomin)
Drug: Placebo — Placebo to incobotulinumtoxinA (Xeomin) powder for solution for injection dose (Main Period only): one injection session of solution, prepared by reconstitution of powder with 0.9% Sodium chloride (NaCl), placebo volume corresponding to up to 50 Units per eye; Mode of administration: intramuscular injection
  Arms: Placebo

SUMMARY:
Patients received one injection with incobotulinumtoxinA (Xeomin) or placebo at baseline. Thereafter, all patients who entered the Open-Label Extension Period (OLEX) received up to five injection sessions of incobotulinumtoxinA (Xeomin) during the OLEX period.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female pretreated outpatients between ages 18 and 80 years (inclusive)
* A clinical diagnosis of bilateral blepharospasm (BEB) characterized by spontaneous, spasmodic, intermittent or persistent involuntary contractions of the orbicular oculi muscles
* A need for injection of Botulinum toxin (defined by a Jankovic Rating Scale (JRS) severity subscore >= 2)
* On a stable dose of other medications (if any) used for focal dystonia treatment (e.g. anticholinergics and benzodiazepines) for at least 3 months prior to and expected throughout the Main Period
* Source documentation of the last two consecutive injection sessions with BOTOX® and a stable satisfactory therapeutic response directly prior to trial entry
* At least 10 weeks must have been passed between the last injection with BOTOX® for BEB and Baseline

Main Exclusion Criteria:

* Atypical variant of BEB caused by inhibition of levator palpebrae muscle
* Myotomy or denervation surgery in the affected muscles (e.g. peripheral denervation and/or spinal cord stimulation)
* The previous two injections with BOTOX® with more than 50 Units per eye
* Hypersensitivity to human serum albumin, sucrose, or Botulinum toxin A
* Neuroleptic induced blepharospasm
* Diagnosis of myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other significant neuromuscular disease which might interfere with the trial
* Treatment with Botulinum toxins for any indication other than BEB within 4 months prior to Baseline and during the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2006-10; Primary Completion 2008-04 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Jankovic, Prof., Study Chair — Houston, Texas
Locations (2):
- Baylor College of Medicine, Houston, Texas, United States
- David King, MD - Private Practice, Halifax, Nova Scotia, Canada

REFERENCES:
- [Result] Jankovic J, Comella C, Hanschmann A, Grafe S. Efficacy and safety of incobotulinumtoxinA (NT 201, Xeomin) in the treatment of blepharospasm-a randomized trial. Mov Disord. 2011 Jul;26(8):1521-8. doi: 10.1002/mds.23658. Epub 2011 Apr 22. PMID 21520284
- [Result] Truong DD, Gollomp SM, Jankovic J, LeWitt PA, Marx M, Hanschmann A, Fernandez HH; Xeomin US Blepharospasm Study Group. Sustained efficacy and safety of repeated incobotulinumtoxinA (Xeomin((R))) injections in blepharospasm. J Neural Transm (Vienna). 2013 Sep;120(9):1345-53. doi: 10.1007/s00702-013-0998-9. Epub 2013 Feb 23. PMID 23435927

RESULTS

PARTICIPANT FLOW:
Groups:
- incobotulinumtoxinA (Xeomin): incobotulinumtoxinA (Xeomin) (active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection
- Placebo: Placebo to incobotulinumtoxinA (Xeomin) powder for solution for injection Dose (Main Period only): one injection session of solution, prepared by reconstitution of powder with 0.9% NaCl;Mode of administration: intramuscular injection
Period: Main Period - 6 to 20 Weeks
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Started | 75 | 34
Completed | 70 | 32
Not Completed | 5 | 2
Not completed — Withdrawal Criteria Occurred | 4 | 0
Not completed — Consent Withdrawn | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Dosing Error At Visit 2 (Baseline) | 0 | 1
Period: Open-Label Ext. Period - up to 68 Weeks
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Started | 102 | 0 (In the Open-Label Extension Period no placebo treatment arm was given.)
Completed | 82 | 0
Not Completed | 20 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Consent Withdrawn | 6 | 0
Not completed — Withdrawal Criteria Occurred | 4 | 0
Not completed — Lack of Efficacy | 4 | 0
Not completed — Subjects Needed Further Injection | 1 | 0
Not completed — Subject Received Botox Injection | 1 | 0
Not completed — Injection in Wrong Muscle | 1 | 0
Not completed — OLEX Drug Given at Baseline | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo | Total
Number analyzed (Participants) | 75 | 34 | 109
Age Continuous [Mean (Standard Deviation); unit: years] | 61.5 (11.0) | 62.6 (8.7) | 61.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 22 | 71
  Male | 26 | 12 | 38

OUTCOME MEASURES:

1. Primary Outcome: Jankovic Rating Scale (JRS) Change From Baseline in the JRS Severity Subscore at Week 6 After Injection (Assessed by a Blinded Independent Rater)
Description: The Jankovic Rating Scale (JRS) is used for classification of the patient's individual symptoms of blepharospasm and for determination of the therapeutic efficacy of study medication. The JRS sumscore is the sum of the two components of the scale:
  * JRS-Severity score which ranges from 0 (=absence of severity) to 4 (=maximum severity)
  * JRS-Frequency score which ranges from 0 (=no frequency) to 4 (=maximum frequency) The change from baseline was calculated as the score at the corresponding visit minus the baseline score.
Time Frame: Baseline, week 6
Population: Intention to treat population: all participants randomized were included in the primary efficacy analysis; Last Observation Carried Forward (LOCF) imputation technique used for missing values
Measure: Least Squares Mean (Standard Error); unit: Points on a scale
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 75 | 34
Points on a scale | -0.8 (0.13) | 0.2 (0.18)
Statistical Analysis 1: Comparison: incobotulinumtoxinA (Xeomin) vs Placebo; The null hypothesis in the analysis of covariance (ANCOVA) model was the absence of difference in the change from baseline in the JRS severity subscore between incobotulinumtoxinA (Xeomin) and placebo. The ANCOVA model was performed 2-sided (type-I error=5 percent) and change from baseline in the JRS Severity subscore assessed by a blinded Independent Rater as dependent variable. The independent variables were treatment, baseline JRS Severity subscore, gender, age, dose group, and pooled center; Test type: Superiority or Other; p < 0.001, ANCOVA — No type I-error adjustment was necessary in this study; Indepent variables in the model were treatment, baseline JRS-Severity score, gender, age, dose, and pooled center; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-1.4 to -0.5]

2. Secondary Outcome: Jankovic Rating Scale (JRS) Change From Baseline in the JRS Severity Subscore at Week 6 After Injection (Assessed by Subject Diary)
Description: as for outcome 1
Time Frame: Baseline, week 6
Population: Intention to treat population by using the Last Observation Carried Forward (LOCF) imputation technique for missing values
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 67 | 32
Points on a scale | -0.75 (1.24) | 0.16 (1.07)

3. Secondary Outcome: Blepharospasm Disability Index (BSDI) Change From Baseline in the BSDI at Week 6 After Injection
Description: The Blepharospasm Disability Index is a scale for the assessment of impairment of specific activities of daily living caused by blepharospasm. The BSDI consists of six items (driving a vehicle; reading; watching TV; shopping; getting about on foot (walking); doing everyday activities), each ranges from 0 (=no impairment) to 4 (=no longer possible due to illness). The change from baseline was calculated as the score at the corresponding visit minus the baseline score.
Time Frame: Baseline, week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 75 | 34
Points on a scale | -0.4 (0.69) | 0.11 (0.67)

4. Secondary Outcome: Patient Evaluation of Global Response (PEGR) at Final Visit
Description: The PEGR is a descriptive subjective 9-point response scale ranging from "complete abolishment of signs and symptoms" (value=+4) down to "very marked worsening" (value=-4).
Time Frame: Final visit (up to week 20 after injection of the Main Period)
Population: Intention to treat population with missing values imputed by "no effect".
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Number analyzed (Participants) | 75 | 34
Points on a scale | 1.3 (2.09) | -0.6 (2.16)

ADVERSE EVENTS:
Time Frame: All SAEs/AEs during Double-Blind Period After Injection, i.e. up to 6-20 weeks after Main Period injection.
Description: The table of "Other Adverse Events" includes all non-serious AEs. Only results and AEs of the Double-Blind Period are given as the Open-Label Extension Period was a non-controlled study. The investigator asked the patient for AEs systematically at each visit.
Arm/Group | incobotulinumtoxinA (Xeomin) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/74 | 1/34
Other Adverse Events (participants affected / at risk) | 45/74 | 13/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | incobotulinumtoxinA (Xeomin) (N=74) | Placebo (N=34)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | incobotulinumtoxinA (Xeomin) (N=74) | Placebo (N=34)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 0 (0)
Dry eye (Eye disorders) | 14 (16) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 11 (11) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Eyelid ptosis (Eye disorders) | 14 (14) | 2 (2)
Headache (Nervous system disorders) | 7 (7) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2)
Respiratory tract infection (Infections and infestations) | 5 (5) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Vision blurred (Eye disorders) | 4 (4) | 2 (2)
Visual disturbance (Eye disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No results to be published without written agreement by sponsor; manuscripts to be sent to sponsor at least 6 weeks before submission. Sponsor to give written opinion within 30 days. Sponsor is entitled to exert influence on the contents of publications, to postpone publications up to 36 months after end of the study, and to name co-authors. In case of justified doubts of sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.